CLINICAL TRIAL: NCT06623513
Title: A Single-Center, Prospective, Randomized, Controlled, Exploratory Trial Comparing the Efficacy and Safety of Parecoxib vs. Indomethacin in Preventing Post-ERCP Pancreatitis: The PRECISE Trail
Brief Title: Efficacy and Safety of Parecoxib vs. Indomethacin in Preventing Post-ERCP Pancreatitis
Acronym: PRECISE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ge Yu, Attending Physician, Gastroenterology Department, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCTR-2023C01
Record Dates: First submitted 2024-09-27; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Pancreatitis, Acute; Cholangiopancreatography, Endoscopic Retrograde
Keywords: Parecoxib; Indomethacin; Post-ERCP Pancreatitis; Efficacy; Safety
MeSH Terms: conditions — Pancreatitis | interventions — parecoxib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parecoxib Group (Experimental)
  Interventions: Drug: Parecoxib Sodium
- Indomethacin Group (Active Comparator)
  Interventions: Drug: Indomethacin suppository

INTERVENTIONS:
Drug: Parecoxib Sodium — Parecoxib Sodium 40 mg administered intravenously 30 minutes before the ERCP procedure.
  Arms: Parecoxib Group
Drug: Indomethacin suppository — Indomethacin suppository 100 mg administered rectally 30 minutes before the ERCP procedure.
  Arms: Indomethacin Group

SUMMARY:
This study aims to evaluate the efficacy and safety of parecoxib versus indomethacin in preventing post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (PEP). It is a single-center, prospective, randomized, controlled, exploratory trial. Participants will be randomly assigned to receive either parecoxib or indomethacin as a preventive treatment. The primary endpoint is to compare the efficacy of the two drugs in reducing the incidence of PEP. Secondary endpoints include the incidence of moderate to severe PEP and post-ERCP-related adverse events. This study will systematically assess the efficacy and safety of both drugs, providing preliminary data for future larger confirmatory trials.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years.
* Patients scheduled to undergo ERCP for conditions such as common bile duct stones, benign or malignant biliary strictures, cholangitis, suspected biliary tumors, unexplained jaundice, or pancreas divisum.

Exclusion Criteria:

* Previous papillectomy.
* Previous endoscopic sphincterotomy (EST) without planned pancreatic duct intervention.
* Simple biliary stent removal or replacement without planned pancreatic duct intervention.
* Biliary-duodenal fistula, post-biliary-duodenal anastomosis, or post-biliary-jejunal anastomosis.
* Malignant tumor of the pancreatic head.
* Currently or recently (within 1 week) suffering from acute pancreatitis.
* Current or recent (within 1 week) use of NSAIDs.
* Recent (within 2 weeks) or within 4 weeks prior to surgery, gastrointestinal bleeding or peptic ulcers.
* History of significant adverse reactions to NSAIDs.
* Renal insufficiency (creatinine clearance < 30 mL/min).
* Moderate to severe hepatic impairment (Child-Pugh score ≥ 7).
* Severe cardiovascular or cerebrovascular disease.
* Patients with psychiatric disorders.
* Pregnant or breastfeeding patients.
* Patients without a rectum.
* Patients unwilling or unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-ERCP Pancreatitis (PEP) | 24 hours after ERCP procedure.
  The primary outcome is the proportion of patients who develop post-ERCP pancreatitis. PEP is characterized by new or worsened abdominal pain, elevated serum amylase levels (≥3 times the upper normal limit).

SECONDARY OUTCOMES:
Incidence of Moderate to Severe PEP | At discharge (up to 30 days)
  The severity of PEP will be classified according to the Cotton consensus and the revised Atlanta classification.
Incidence of Hyperamylasemia | 3 and 24 hours after ERCP procedure
  Hyperamylasemia is defined as a serum amylase level greater than three times the upper limit of normal, without the onset of new abdominal pain or worsening of existing pain.
Post-Procedure Discomfort Symptoms | Baseline (pre-procedure), 3 hours post-procedure, 6 hours post-procedure, 12 hours post-procedure, 24 hours post-procedure, 48 hours post-procedure, 72 hours post-procedure, and at discharge (up to 30 days)
  Definition: Post-ERCP discomfort symptoms primarily include abdominal pain, nausea, vomiting, sore throat, abdominal bloating, dizziness, and headache. To comprehensively assess the severity of these symptoms, the study will utilize the Symptom Severity Index (SSI) to quantify and analyze patient-reported symptoms.
  Assessment Method: Each symptom will be self-assessed by the patient using the Numeric Rating Scale (NRS), a self-assessment tool, and verified by the study staff. The score ranges from 0 to 10, where 0 represents no symptoms, and 10 represents the most severe symptoms.
  Scoring Weights: The final score for each symptom will be calculated by multiplying the symptom score by its respective weight. The total symptom score will be the sum of all weighted scores, with a maximum score of 100.
Bleeding, Perforation, Cholangitis, Cardiac Adverse Events, Renal Adverse Events | 3 hours post-procedure, 6 hours post-procedure, 12 hours post-procedure, 24 hours post-procedure, 48 hours post-procedure, 72 hours post-procedure, and at discharge (up to 30 days)
  Symptom-driven detection methods will be used to evaluate adverse events. The severity of bleeding, perforation, and cholangitis will be assessed according to the Cotton criteria.

IPD SHARING:
Plan to Share IPD: No